CLINICAL TRIAL: NCT02214797
Title: Dispensing Study to Assess Visual Performance of Prototype Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brien Holden Vision (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CRTC2013-02; ACTRN12614000011684 (Registry Identifier: ANZCTR)
Record Dates: First submitted 2014-08-07; First posted 2014-08-12 (Estimated); Last update posted 2015-06-25 (Estimated); Status verified 2015-06

CONDITIONS: Presbyopia; Refractive Error
Keywords: Presbyopia; Refractive Error; Contact Lenses
MeSH Terms: conditions — Presbyopia; Refractive Errors

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Presbyopic group - Low Add (Other): 40 years and over Add of less than +1.50D
  Control lens : Lotrafilcon B and Senofilcon A
  Test lens: Etafilcon A
  Up to 4 test lens designs will be assessed against commercial control/s in each parallel arm in a randomised cross over fashion. Each lenses will be worn for a week with a minimum 2 day washout period between the lens types. Each lens will require 2 scheduled clinic attendances - a fitting visit and an evaluation visit.
  Interventions: Device: Etafilcon A, Lotrafilcon B , Senofilcon A
- Presbyopic group - Med Add (Other): 40 years and over Add of +1.50D to +1.75D
  Control lens : Lotrafilcon B and Senofilcon A
  Test lens: Etafilcon A
  Up to 4 test lens designs will be assessed against commercial control/s in each parallel arm in a randomised cross over fashion, with a minimum 2 day washout period between the lens types. Each lens assessment will require 2 scheduled clinic attendances - a fitting visit and an evaluation visit.
  Interventions: Device: Etafilcon A, Lotrafilcon B , Senofilcon A
- Presbyopic group - High Add (Other): 40 years and over Add of +2.00D to +2.50D
  Control lens : Lotrafilcon B and Senofilcon A
  Test lens: Etafilcon A
  Up to 4 test lens designs will be assessed against commercial control/s in each parallel arm in a randomised cross over fashion, with a minimum 2 day washout period between the lens types. Each lens assessment will require 2 scheduled clinic attendances - a fitting visit and an evaluation visit.
  Interventions: Device: Etafilcon A, Lotrafilcon B , Senofilcon A
- Non-presbyopic group (Other): 18 to 39 years old No Add
  Control lens : Lotrafilcon B and Etafilcon A
  Test lens: Etafilcon A
  Up to 4 test lens designs will be assessed against commercial control/s in each parallel arm in a randomised cross over fashion, with a minimum 2 day washout period between the lens types. Each lens assessment will require 2 scheduled clinic attendances - a fitting visit and an evaluation visit.
  Interventions: Device: Etafilcon A, Lotrafilcon B , Senofilcon A

INTERVENTIONS:
Device: Etafilcon A, Lotrafilcon B , Senofilcon A
  Other Names: Control lenses; Non-presbyopic group; Brand name: Air Optix® Aqua , Acuvue® 1-Day Moist; Lens material: Lotrafilcon B , Etafilcon A; Presbyopic group; Brand name: Air Optix® Multifocal, Acuvue® Oasys for Presbyopia; Lens material Lotrafilcon B, Senofilcon A; Test lens; Brand name: Iteration X; Lens material: Etafilcon A

SUMMARY:
The aim of this study is to assess visual performance of prototype soft contact lens designs compared to commercially available contact lenses over one-week of lens wear.

DETAILED DESCRIPTION:
Prospective, participant-masked, multiple arm, crossover dispensing clinical trial where participants will wear prototype (test) and commercial (control) lenses bilaterally. Participants will be stratified based on their refractive error into either presbyopic or non-presbyopic group. Each of the stratified group will have a maximum of 4 parallel arms. Up to 4 test lens designs will be assessed against the control/s in each parallel arm in a randomized cross over fashion, with a minimum 2 day washout period between the lens types. Each lens assessment will require 2 scheduled clinic attendances - a fitting visit and an evaluation visit.

ELIGIBILITY:
Inclusion Criteria:

* Able to read and comprehend English and give informed consent as demonstrated by signing a record of informed consent
* Be at least 18 years old, male or female
* Willing to comply with the wearing and clinical trial visit schedule as directed by the Investigator
* Have ocular health findings considered to be "normal" and which would not prevent the participant from safely wearing contact lenses
* Correctable to at least 6/12 (20/40) or better in each eye with contact lenses
* Be willing to not wear contact lenses for a minimum of 2 days before each stage of the clinical trial (after informed consent)

Exclusion Criteria:

* Any pre-existing ocular irritation, injury or condition (including infection or disease) of the cornea, conjunctiva or eyelids that would preclude contact lens fitting and safe wearing of contact lenses
* Any systemic disease that adversely affects ocular health e.g. diabetes, Graves disease, and auto immune diseases such as ankylosing spondylitis, multiple sclerosis, Sjögrens syndrome and systemic lupus erythematosus. Conditions such as systemic hypertension and arthritis do not automatically exclude prospective participants
* Use of or a need for concurrent category S3 and above ocular medication at enrolment and/or during the clinical trial
* Use of or a need for any systemic medication or topical medications which may alter normal ocular findings / are known to affect a participant's ocular health / physiology or contact lens performance either in an adverse or beneficial manner at enrolment and/or during the clinical trial NB: Systemic antihistamines are allowed on an "as needed basis", provided they are not used prophylactically during the trial and at least 24 hours before the clinical trial product is used
* Eye surgery within 12 weeks immediately prior to enrolment for this trial.
* Previous corneal refractive surgery
* Contraindications to contact lens wear
* Known allergy or intolerance to ingredients in any of the clinical trial products

The Investigator may, at his/her discretion, exclude anyone who they believe may not be able to fulfil the clinical trial requirements or it is believed to be in the participant's best interests

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2014-09; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Change in visual performance over 1-week lens wear | after about 20 minutes of lens wear and after about 1 week of lens wear
  Visual Acuity Visual acuity will be recorded on an interval scale. Data will be summarised as means ± standard deviations. No transformation is likely to be required. Visual acuity will be compared between test and control lens types and time across 1 week. Interactions will be tested and, if present, the significance of lens types will be determined at each time point and over time for each lens type. Visual acuity will be analysed using linear mixed model with subject random intercepts and / or paired t-test.

SECONDARY OUTCOMES:
Change in subjective response over 1-week of lens wear | After about 40 mins of lens wear and after 2 days, 4 days and 1 week of lens wear
  Subjective ratings Questionnaire Subjective ratings will be recorded on a scale of 1 to 10 on steps of 1. Data will be summarised as means ± standard deviations. No transformation is likely to be required. Subjective ratings will be compared between test and control lens types and time across 1 week. Interactions will be tested and, if present, the significance of lens type will be determined at each time point and over time for each lens type. Subjective ratings will be analysed using linear mixed model with subject random intercepts and / or paired t-test.

CONTACTS AND LOCATIONS:
Overall Officials: Jiyoon Chung, BOptom, Principal Investigator — Brien Holden Vision Institute
Locations (1):
- Brien Holden Vision Institue, Clinical Research Trials Center, Sydney, New South Wales, Australia

REFERENCES:
- [Background] Young G, Veys J, Pritchard N, Coleman S. A multi-centre study of lapsed contact lens wearers. Ophthalmic Physiol Opt. 2002 Nov;22(6):516-27. doi: 10.1046/j.1475-1313.2002.00066.x. PMID 12477016
- [Background] Stapleton F, Keay L, Edwards K, Naduvilath T, Dart JK, Brian G, Holden BA. The incidence of contact lens-related microbial keratitis in Australia. Ophthalmology. 2008 Oct;115(10):1655-62. doi: 10.1016/j.ophtha.2008.04.002. Epub 2008 Jun 5. PMID 18538404
- [Derived] Jong M, Tilia D, Sha J, Diec J, Thomas V, Bakaraju RC. The Relationship between Visual Acuity, Subjective Vision, and Willingness to Purchase Simultaneous-image Contact Lenses. Optom Vis Sci. 2019 Apr;96(4):283-290. doi: 10.1097/OPX.0000000000001359. PMID 30907859